CLINICAL TRIAL: NCT07054099
Title: A Phase III, Double-blind, Randomized, Multicenter, Multinational, Active-controlled, Non-inferiority Study to Evaluate Immunogenicity and Safety After the First and Second Doses of MG1111 (BARYCELA Inj.) in Healthy Children Aged 12 Months to 12 Years
Brief Title: A Study to Evaluate Immunogenicity and Safety After the First and Second Doses of MG1111 (BARYCELA Inj.) in Healthy Children Aged 12 Months to 12 Years
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MG1111_VAR2D_P0304
Record Dates: First submitted 2025-07-07; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Varicella (Chickenpox); Chickenpox Vaccine
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG1111 (Barycela inj.) (Experimental)
  Interventions: Biological: MG1111 (Barycela inj.)
- Varivax™ (Active Comparator)
  Interventions: Biological: VARIVAX™

INTERVENTIONS:
Biological: MG1111 (Barycela inj.) — MG1111 (Barycela inj.)
  Arms: MG1111 (Barycela inj.)
Biological: VARIVAX™ — Varivax™
  Arms: Varivax™

SUMMARY:
This clinical study aims to evaluate the safety and immune response of MG1111, in healthy children compared to VARIVAX. The study will follow participants for 42 days after receiving two doses, with additional follow-ups for up to 10 years to monitor varicella infection.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 12 months to 12 years of age, inclusive, at the time of signing the informed consent or assent.
* Participant is overtly healthy as determined by the investigator

Exclusion Criteria:

* Participants with a history of exposure to varicella through contact with a varicella patient at home, school, or childcare facility within 4 weeks before Screening
* Participants with a history of varicella infection and varicella vaccine, either licensed or investigational, and either standalone or any combination, such as MMRV
* Participants with acute moderate or severe infection with or without fever at the time of dosing
* Participants who have had any suspected allergy symptoms, such as systemic rash, during the 72 hours before each administration of investigational product

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 474 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieved seroconversion at 42 days after second vaccination | 42 days after second vaccination

SECONDARY OUTCOMES:
Percentage of participants reporting local and systemic solicited adverse events during the first 7 days after each vaccination with MG1111 or VARIVAX | 7 days after each vaccination
Percentage of participants reporting unsolicited adverse events during the first 42 days after each vaccination with MG1111 or VARIVAX | 42 days after each vaccination
Percentage of participants reporting serious adverse events until 6 months after second vaccination with MG1111 or VARIVAX | 6 months after second vaccination